CLINICAL TRIAL: NCT05833451
Title: Is Reiki Effective In Coping With the Symptoms Experienced by Patients Undergoing Hemodialysis?: Single-Blind Randomized Controlled Trial
Brief Title: Reiki in Symptom Management of Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Ulviye Özcan Yüce, PhD., Assist. Prof., Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/02/12-E.54558
Record Dates: First submitted 2023-03-29; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Renal Dialysis
Keywords: nursing; hemodialysis; Reiki; urea; hemodialysis symptoms
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): The participants in the Reiki group (n=32) were given Reiki remotely for 60 minutes by two certified practitioners who completed the second level Reiki training with a Master degree Reiki instructor according to the Usui method.
  Interventions: Other: Reiki
- Control (No Intervention): No intervention was made in the control group (n=32).

INTERVENTIONS:
Other: Reiki — Reiki, one of integrative practices, is an energy therapy involving the use of energy that flows naturally from the hands of the practitioner to strengthen the body's ability to heal itself in order to increase well-being. Reiki improves well-being in many areas, ensures that blood and lymph circulation is maintained properly, regulates blood pressure and pulse rate by stimulating the autonomic nervous system, increases comfort, reduces depression and anxiety levels. In this way, Reiki facilitates physical and mental relaxation and promotes health
  Arms: Reiki

SUMMARY:
This study aims to investigate the effect of Reiki applied to individuals receiving hemodialysis treatment on hemodialysis-related symptoms and hematological indicators.

DETAILED DESCRIPTION:
The study has a pretest-posttest randomized controlled design and it was carried out between March and July 2022 with 64 patients over the age of 18 who received hemodialysis treatment for at least 15 days in the dialysis unit of state hospitals in two different cities. Data were collected using the Patient Information Form, the Dialysis Symptom Index (DSI), and the follow-up chart including erythrocyte (RBC), hemoglobin (HGB), hematocrit (HCT), serum urea, creatinine, sodium (Na), potassium (K), phosphorus (P), and calcium (Ca) values. While the distance Reiki intervention was applied to each of the patients in the Reiki group for 60 minutes, no intervention was made in the control group. One week after the intervention, the DSI was re-administered to the patients in the posttest, and hematology and biochemistry results were recorded.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years of age,
* To have received hemodialysis treatment for at least 15 days,
* To volunteer to participate in the study,
* To be able to answer the given forms and questionnaires

Exclusion Criteria:

* To be a Reiki practitioner or trainer,
* To have attended any energy therapy session before,
* Using other complementary and integrative medicine practices at the time of the application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline Dialysis Symptom Index at a week | Within 1 hour of first admission. -A week later
  The Dialysis Symptom Index was used to investigate the therapeutic effect of Reiki on hemodialysis-related symptoms. The index consists of 30 items to evaluate physical and emotional symptoms and the severity of these symptoms. Participants are asked to define the presence of each symptom they experienced in the last week as Yes or No, and they are also report how much symptoms they experience affect them on a five-point Likert type scale (1 = not at all bothersome, 5 = very much bothersome). The lowest score to be obtained from the index is 0, the highest score is 150, and higher scores indicate more dialysis symptoms. In order to reach the Primary Outcome Measure, it was aimed that the Dialysis Symptom Index total scores of the individuals in the intervention group were lower in the final measurement than in the first measurement.

SECONDARY OUTCOMES:
Change from Sodium values at a week | Within one week of first application
  In this section there is Sodium value required for eliminating fluid-electrolyte imbalances. The observed sodium is expected to be 136 -144 mmol/L.
Change from Potassium values at a week | Within one week of first application
  In this section there is Potassium value required for eliminating fluid-electrolyte imbalances. The observed sodium is expected to be 3.7 - 5.1 mmol/L
Change from Calcium values at a week | Within one week of first application
  In this section there is Calcium value required for eliminating fluid-electrolyte imbalances. The observed Calcium is expected to be 8.5 -10.2 mg/dL
Change from Chloride values at a week | Within one week of first application
  In this section there is Chloride value required for eliminating fluid-electrolyte imbalances. The observed Chloride is expected to be 97 - 105 mmol/L
Change from Magnesium values at a week | Within one week of first application
  In this section there is Magnesium value required for eliminating fluid-electrolyte imbalances. The observed Magnesium is expected to be 1.7- 2.2 mg/dL
Change from Phosphate values at a week | Within one week of first application
  In this section there is Phosphate value required for eliminating fluid-electrolyte imbalances. The observed Phosphate is expected to be 2.5- 4.8 mg/dL
Change from urea values at a week | Within one week of first application
  In this section there is urea value required for eliminating fluid-electrolyte imbalances. The observed urea is expected to be 1.8 to 7.1 mmol
Change from Hemoglobin values at a week | Within one week of first application
  In this section there is Hemoglobin value required for preventing anemia. The observed Hemoglobin is expected to be Male (ages 15+): 13.0 - 17.0 g/dL; Female (ages 15+): 11.5 - 15.5 g/dL
Change from Hematocrit values at a week | Within one week of first application
  This section contains the Hematocrit value, which should be in the appropriate range to prevent fluid imbalance and anemia. The observed Hematocrit is expected to be Male: 40 - 55%; Female: 36 - 48%

CONTACTS AND LOCATIONS:
Locations (1):
- Osmaniye Korkut Ata University, Osmaniye, Turkey (Türkiye)

REFERENCES:
- [Background] Duranton F, Cohen G, De Smet R, Rodriguez M, Jankowski J, Vanholder R, Argiles A; European Uremic Toxin Work Group. Normal and pathologic concentrations of uremic toxins. J Am Soc Nephrol. 2012 Jul;23(7):1258-70. doi: 10.1681/ASN.2011121175. Epub 2012 May 24. PMID 22626821
- [Background] Lu PH, Yu MC, Wei MJ, Kuo KL. The Therapeutic Strategies for Uremic Toxins Control in Chronic Kidney Disease. Toxins (Basel). 2021 Aug 17;13(8):573. doi: 10.3390/toxins13080573. PMID 34437444
- [Background] Yu IC, Fang JT, Tsai YF. Exploring demands of hemodialysis patients in Taiwan: A two-step cluster analysis. PLoS One. 2020 Feb 7;15(2):e0228259. doi: 10.1371/journal.pone.0228259. eCollection 2020. PMID 32032397
- [Background] Zarantonello D, Rhee CM, Kalantar-Zadeh K, Brunori G. Novel conservative management of chronic kidney disease via dialysis-free interventions. Curr Opin Nephrol Hypertens. 2021 Jan;30(1):97-107. doi: 10.1097/MNH.0000000000000670. PMID 33186220
- [Background] Kalantar-Zadeh K, Jafar TH, Nitsch D, Neuen BL, Perkovic V. Chronic kidney disease. Lancet. 2021 Aug 28;398(10302):786-802. doi: 10.1016/S0140-6736(21)00519-5. Epub 2021 Jun 24. PMID 34175022
- [Background] Vanholder RC, Eloot S, Glorieux GL. Future Avenues to Decrease Uremic Toxin Concentration. Am J Kidney Dis. 2016 Apr;67(4):664-76. doi: 10.1053/j.ajkd.2015.08.029. Epub 2015 Oct 21. PMID 26500179
- [Background] Li PK, Garcia-Garcia G, Lui SF, Andreoli S, Fung WW, Hradsky A, Kumaraswami L, Liakopoulos V, Rakhimova Z, Saadi G, Strani L, Ulasi I, Kalantar-Zadeh K. Kidney health for everyone everywhere - from prevention to detection and equitable access to care. Clin Nephrol. 2020 Mar;93(3):111-122. doi: 10.5414/CNWKDEditorial. PMID 32017699
- [Background] Komenda P, Ferguson TW, Macdonald K, Rigatto C, Koolage C, Sood MM, Tangri N. Cost-effectiveness of primary screening for CKD: a systematic review. Am J Kidney Dis. 2014 May;63(5):789-97. doi: 10.1053/j.ajkd.2013.12.012. Epub 2014 Feb 12. PMID 24529536
- [Background] Weisbord SD, Fried LF, Arnold RM, Rotondi AJ, Fine MJ, Levenson DJ, Switzer GE. Development of a symptom assessment instrument for chronic hemodialysis patients: the Dialysis Symptom Index. J Pain Symptom Manage. 2004 Mar;27(3):226-40. doi: 10.1016/j.jpainsymman.2003.07.004. PMID 15010101
- [Background] Daniel P. Wirth, R. J. Chang, W. S. Eidelman & J. B. Paxton, Hematological Indicators of Complementary Healing Intervention, Complementary Therapies in Medicine 4 (996), pp. 4-20.
- [Background] Önsöz HB, Usta Yeşilbalkan Ö. Reliability and validity of the Turkish version of the dialysis symptom index in chronic hemodialysis patients. Turkish Nephrology, Dialysis and Transplantation Journal 2013; 22(1): 60-67
- [Background] Dyer NL, Baldwin AL, Rand WL. A Large-Scale Effectiveness Trial of Reiki for Physical and Psychological Health. J Altern Complement Med. 2019 Dec;25(12):1156-1162. doi: 10.1089/acm.2019.0022. Epub 2019 Oct 22. PMID 31638407
- [Background] Zins S, Hooke MC, Gross CR. Reiki for Pain During Hemodialysis: A Feasibility and Instrument Evaluation Study. J Holist Nurs. 2019 Jun;37(2):148-162. doi: 10.1177/0898010118797195. Epub 2018 Aug 31. PMID 30170509
- [Background] Muhith A, Hidayaah N, Faizah I, Sari, RY, Hartadi H. The Effect of Reiki Therapy on Posttraumatic Growth (Ptg) Among Chronic Renal Failure Patients Through Hemodialysis. Nurse and Health: Journal Keperawatan. 2021, 10(2): 190-200. http://ejournal-kertacendekia.id/index.php/nhjk/index